CLINICAL TRIAL: NCT02576977
Title: A Phase III Study of Pomalidomide and Low Dose Dexamethasone With or Without Pembrolizumab (MK3475) in Refractory or Relapsed and Refractory Multiple Myeloma (rrMM) (KEYNOTE 183)
Brief Title: Study of Pomalidomide and Low Dose Dexamethasone With or Without Pembrolizumab (MK-3475) in Refractory or Relapsed and Refractory Multiple Myeloma (rrMM) (MK-3475-183/KEYNOTE-183)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated early due to business reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-183; 2015-002509-13 (EudraCT Number); 163146 (Registry Identifier: JAPAN-CTI); MK-3475-183 (Other: Merck Protocol Number); KEYNOTE-183 (Other: Merck)
Record Dates: First submitted 2015-10-14; First posted 2015-10-15 (Estimated); Results first posted 2019-08-02 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Multiple Myeloma
Keywords: PDL1; PD1; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — pembrolizumab; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab+Pomalidomide+Dexamethasone (Experimental): Participants receive pembrolizumab 200 mg intravenously (IV) on Day 1 every 3 weeks (Q3W) PLUS pomalidomide 4 mg orally (PO) on Days 1 to 21 of each 28-day cycle PLUS dexamethasone 40 mg PO on Days 1, 8, 15 and 22 of each 28-day cycle.
  Interventions: Biological: Pembrolizumab; Drug: Pomalidomide; Drug: Dexamethasone
- Pomalidomide+Dexamethasone (Active Comparator): Participants receive pomalidomide 4 mg PO on Days 1 to 21 of each 28-day cycle PLUS dexamethasone 40 mg PO on Days 1, 8, 15 and 22 of each 28-day cycle.
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Biological: Pembrolizumab — pembrolizumab 200 mg IV infusion
  Other Names: KEYTRUDA®; MK-3475; SCH 9000475
  Arms: Pembrolizumab+Pomalidomide+Dexamethasone
Drug: Pomalidomide — pomalidomide 4 mg capsules
  Other Names: POMALYST®
Drug: Dexamethasone — dexamethasone 40 mg tablets

SUMMARY:
The purpose of this study is to compare the efficacy of pomalidomide and low dose dexamethasone with pembrolizumab (MK-3475) to that of pomalidomide and low dose dexamethasone without pembrolizumab in terms of Progression-Free Survival (PFS) in participants with refractory or relapsed and refractory multiple myeloma (rrMM) who have undergone at least 2 lines of prior treatment. The study's 2 primary hypotheses are: 1. Pembrolizumab in combination with pomalidomide and low dose dexamethasone prolongs PFS as assessed by Clinical Adjudication Committee (CAC) blinded central review using International Myeloma Working Group Criteria for Response Assessment in Multiple Myeloma (IMWG) criteria compared to treatment with pomalidomide and low dose dexamethasone standard of care (SOC) alone. 2. Pembrolizumab in combination with pomalidomide and low dose dexamethasone prolongs OS compared to treatment with pomalidomide and low dose dexamethasone (SOC) alone.

ELIGIBILITY:
Inclusion Criteria:

* Has a confirmed diagnosis of active multiple myeloma and measurable disease
* Must have undergone prior treatment with ≥2 treatment lines of anti-myeloma therapy and must have failed last line of treatment (refractory to last line of treatment)
* Prior anti-myeloma treatments must have included an immunomodulatory drug (IMiD) AND proteasome inhibitor alone or in combination and participant must have failed therapy with an IMiD OR proteasome inhibitor
* Has performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Female participants of childbearing potential must have 2 negative urine human chorionic gonadotropin tests within 10 to 14 days and within 24 hours prior to receiving study medication
* Female participants of childbearing potential and male participants must agree to use adequate contraception 28 days prior to study start and continuing for up to 28 days after the last dose of pomalidomide (or 120 days after the last dose of pembrolizumab)

Exclusion Criteria:

* Has had prior anti-myeloma therapy within 2 weeks prior to study start and has not recovered (i.e., ≤ Grade 1 or at Baseline) from adverse events due to a previously administered agent
* Has undergone prior allogeneic hematopoietic stem cell transplantation within the last 5 years. (Participants who have had a transplant greater than 5 years ago are eligible as long as there are no symptoms of Graft versus Host Disease [GVHD]).
* Has received autologous stem cell transplant (auto-SCT) within 12 weeks before the first infusion or is planning for or is eligible for auto-SCT
* Has received previous therapy with pomalidomide
* Has peripheral neuropathy ≥ Grade 2
* Has a known additional malignancy that is progressing or requires active treatment within the last 5 years (except for basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy)
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has received prior therapy with an anti-programmed cell death 1 receptor (anti-PD-1), antiprogrammed death-ligand 1 (anti-PD-L1), anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways)
* Is pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2020-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Liao JJZ, Farooqui MZH, Marinello P, Hartzel J, Anderson K, Ma J, Gause CK. Using artificial intelligence tools in answering important clinical questions: The KEYNOTE-183 multiple myeloma experience. Contemp Clin Trials. 2020 Dec;99:106179. doi: 10.1016/j.cct.2020.106179. Epub 2020 Oct 18. PMID 33086159
- [Derived] Mateos MV, Blacklock H, Schjesvold F, Oriol A, Simpson D, George A, Goldschmidt H, Larocca A, Chanan-Khan A, Sherbenou D, Avivi I, Benyamini N, Iida S, Matsumoto M, Suzuki K, Ribrag V, Usmani SZ, Jagannath S, Ocio EM, Rodriguez-Otero P, San Miguel J, Kher U, Farooqui M, Liao J, Marinello P, Lonial S; KEYNOTE-183 Investigators. Pembrolizumab plus pomalidomide and dexamethasone for patients with relapsed or refractory multiple myeloma (KEYNOTE-183): a randomised, open-label, phase 3 trial. Lancet Haematol. 2019 Sep;6(9):e459-e469. doi: 10.1016/S2352-3026(19)30110-3. Epub 2019 Jul 18. PMID 31327687
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject Disposition as per database cutoff date of August 3, 2020.
Pre-assignment Details: Note: For administrative reasons (a noncompliant site), one participant in the SOC arm was recorded as "Ongoing in Trial" in the CSR Disposition Table and "Final Disposition Unknown" here.
Groups:
- Standard of Care (SOC) Pomalidomide+Dexamethasone: Participants receive pomalidomide 4 mg PO on Days 1 to 21 of each 28-day cycle PLUS dexamethasone 40 mg PO on Days 1, 8, 15 and 22 of each 28-day cycle.
Period: Overall Study
Arm/Group | Pembrolizumab+Pomalidomide+Dexamethasone | Standard of Care (SOC) Pomalidomide+Dexamethasone
Started | 126 | 125
Treated | 122 | 123
Completed | 0 | 0
Not Completed | 126 | 125
Not completed — Adverse Event | 13 | 2
Not completed — Death | 73 | 60
Not completed — Screen failure | 1 | 0
Not completed — Study Terminated at Selected Sites | 27 | 50
Not completed — Withdrawal by Subject | 11 | 11
Not completed — Final Disposition Unknown | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Progressive Disease | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab+Pomalidomide+Dexamethasone | Standard of Care (SOC) Pomalidomide+Dexamethasone | Total
Number analyzed (Participants) | 126 | 125 | 251
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.5 (9.3) | 66.4 (10.0) | 65.9 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 46 | 94
  Male | 78 | 79 | 157
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 5 | 13
  Not Hispanic or Latino | 110 | 117 | 227
  Unknown or Not Reported | 8 | 3 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 17 | 12 | 29
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 10 | 14 | 24
  White | 92 | 95 | 187
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 4 | 1 | 5
Disease Status (Refractory vs. Sensitive to Lenalidomide) [Count of Participants; unit: Participants]
  Refractory to Lenalidomide | 108 | 108 | 216
  Sensitive to Lenalidomide | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Assessed by Clinical Adjudication Committee (CAC) Blinded Central Review According to the International Myeloma Working Group (IMWG) Response Criteria
Description: Progression free survival was defined as the time from randomization to the first documented disease progression, or death due to any cause, whichever occurred first. PFS was assessed by CAC blinded central review according to the IMWG criteria based on the development of new bone lesions or soft tissue plasmacytomas or on a definite increase in the size of existing bone lesions or soft tissue plasmacytomas. Median PFS was calculated from the product-limit (Kaplan-Meier) method for censored data. The database cutoff date was July 9, 2018.
Time Frame: Up to approximately 30 months
Population: The analysis population included all randomized participants. Participants were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Pomalidomide+Dexamethasone | Standard of Care (SOC) Pomalidomide+Dexamethasone
Number analyzed (Participants) | 126 | 125
Months | 5.7 [4.5 to 7.5] | 7.4 [5.6 to 11.5]
Statistical Analysis 1: Comparison: Pembrolizumab+Pomalidomide+Dexamethasone vs Standard of Care (SOC) Pomalidomide+Dexamethasone; Test type: Superiority; p = 0.99324, Log Rank; One-sided p-value based on Stratified log-rank test; Hazard Ratio (HR) = 1.50, 95% CI 2-sided [1.08 to 2.08] — Based on Cox regression model with treatment as a covariate stratified by disease status (refractory vs. sensitive to Lenalidomide) and Lines of previous treatments (two vs. three or more)

2. Primary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. Median overall survival was calculated from the product-limit (Kaplan-Meier) method for censored data. The database cutoff date was August 3, 2020.
Time Frame: Up to approximately 54 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Pomalidomide+Dexamethasone | Standard of Care (SOC) Pomalidomide+Dexamethasone
Number analyzed (Participants) | 126 | 125
Months | 21.0 [14.2 to 29.1] | 39.6 [28.5 to NA] — OS upper limit was not reached due to an insufficient number of deaths.
Statistical Analysis 1: Comparison: Pembrolizumab+Pomalidomide+Dexamethasone vs Standard of Care (SOC) Pomalidomide+Dexamethasone; Test type: Superiority; p = 0.99989, Log Rank; One-sided p-value based on Stratified log-rank test; Hazard Ratio (HR) = 1.84, 95% CI 2-sided [1.32 to 2.55]; The Hazard Ratio and 95% confidence intervals were based on Cox regression model with treatment as a covariate stratified by disease status (refractory vs. sensitive to Lenalidomide) and Lines of previous treatments (two vs. three or more)

3. Secondary Outcome: Overall Response Rate (ORR) Evaluated According to the IMWG Response Criteria by CAC Blinded Central Review
Description: ORR was defined as the percentage of the participants in the analysis population who achieved at least a partial response (stringent complete response [sCR]+complete response [CR]+very good partial response [VGPR]+partial response [PR]) according to the IMWG. CR = negative immunofixation of serum and urine AND disappearance of any soft tissue plasmacytomas AND <5% plasmacytomas in the bone marrow; sCR=stringent complete response, CR as above PLUS normal serum free light-chain (FLC) assay ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence; VGPR = serum and urine M-component detectable by immunofixation but not on electrophoresis OR ≥ 90% reduction in serum M-component plus urine M-component <100 mg/24 hr; PR = ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 hours. The database cutoff date was July 9, 2018.
Time Frame: Up to approximately 30 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab+Pomalidomide+Dexamethasone | Standard of Care (SOC) Pomalidomide+Dexamethasone
Number analyzed (Participants) | 126 | 125
Percentage of participants | 37.3 [28.9 to 46.4] | 42.4 [33.6 to 51.6]
Statistical Analysis 1: Comparison: Pembrolizumab+Pomalidomide+Dexamethasone vs Standard of Care (SOC) Pomalidomide+Dexamethasone; Test type: Superiority; p = 0.79921, Miettinen & Nurminen method; Difference in % vs. SOC = -5.2, 95% CI 2-sided [-17.1 to 6.9]; Based on Miettinen & Nurminen method stratified by disease status (refractory vs. sensitive to Lenalidomide) and Lines of previous treatments (two vs. three or more); If there were no participants in one of the treatment groups involved in a comparison for a particular stratum, then that stratum was excluded from the treatment comparison

4. Secondary Outcome: Participants Experiencing One or More Adverse Events (AEs)
Description: An adverse event (AE) was defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it was considered related to the medical treatment or procedure, that occurred during the course of the study. Database cutoff was August 3, 2020.
Time Frame: Up to approximately 54 months
Population: The analysis population consisted of all randomized participants who received at least one dose of study treatment. Participants were included in the treatment group corresponding to the study treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab+Pomalidomide+Dexamethasone | Standard of Care (SOC) Pomalidomide+Dexamethasone
Number analyzed (Participants) | 122 | 123
Participants | 122 | 119

5. Secondary Outcome: Participants Discontinuing Study Investigational Product Due to an AE
Description: An adverse event was defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it was considered related to the medical treatment or procedure, that occurred during the course of the study. Database cutoff was August 3, 2020.
Time Frame: Up to approximately 54 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab+Pomalidomide+Dexamethasone | Standard of Care (SOC) Pomalidomide+Dexamethasone
Number analyzed (Participants) | 122 | 123
Participants | 26 | 10

6. Secondary Outcome: Disease Control Rate (DCR) Evaluated According to the IMWG Response Criteria by CAC Blinded Central Review
Description: Disease control rate was the percentage of participants who achieved confirmed sCR, CR, VGPR, PR, minimal response (MR) or have demonstrated stable disease (SD) for at least 12 weeks prior to any evidence of progression. PD was development of or an increase in the size of bone lesions or soft tissue plasmacytomas. CR = negative immunofixation of serum and urine AND disappearance of any soft tissue plasmacytomas AND <5% plasmacytomas in the bone marrow; sCR=stringent complete response, CR as above PLUS normal serum FLC assay ratio and absence of clonal cells in bone marrow by immunohistochemistry/fluorescence; VGPR = serum and urine M-component detectable by immunofixation but not on electrophoresis OR ≥ 90% reduction in serum M-component plus urine M-component <100 mg/24 hr; PR = ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 hours. The data cutoff date was July 9, 2018.
Time Frame: Up to approximately 30 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab+Pomalidomide+Dexamethasone | Standard of Care (SOC) Pomalidomide+Dexamethasone
Number analyzed (Participants) | 126 | 125
Percentage of participants | 88.1 [81.1 to 93.2] | 84.8 [77.3 to 90.6]

7. Secondary Outcome: Second Progression Free Survival (PFS2)
Description: PFS2 was defined as the time from randomization to subsequent disease progression after initiation of new anti-cancer therapy, or death from any cause, whichever occurred first, by investigator assessment. As a result of a full clinical hold by FDA that led to discontinuation of study enrollment, no data was collected for analysis of PFS2.
Time Frame: Up to approximately 30 months
Population: The analysis population was to include all randomized participants. Study treatment was terminated early and no data was collected for analysis of PFS2.
Arm/Group | Pembrolizumab+Pomalidomide+Dexamethasone | Standard of Care (SOC) Pomalidomide+Dexamethasone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 54 months
Description: The analysis population for all-cause mortality was all randomized participants and for adverse events was the treated participants. Per protocol, disease progression of cancer under study was not considered an adverse event (AE) unless considered related to study treatment, therefore, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study treatment are excluded as AEs. The database cutoff date was August 3, 2020.
Arm/Group | Pembrolizumab+Pomalidomide+Dexamethasone | Standard of Care (SOC) Pomalidomide+Dexamethasone
All-Cause Mortality (participants affected / at risk) | 86/126 | 64/125
Serious Adverse Events (participants affected / at risk) | 79/122 | 57/123
Other Adverse Events (participants affected / at risk) | 115/122 | 114/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab+Pomalidomide+Dexamethasone (N=122) | Standard of Care (SOC) Pomalidomide+Dexamethasone (N=123)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 4 (5)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (2) | 0 (0)
Pericardial haemorrhage (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 5 (5)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Genital herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (4) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 2 (2) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 23 (29) | 17 (21)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia parainfluenzae viral (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 3 (3)
Septic shock (Infections and infestations) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Basosquamous carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
IIIrd nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 4 (4)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 2 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Steroid diabetes (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab+Pomalidomide+Dexamethasone (N=122) | Standard of Care (SOC) Pomalidomide+Dexamethasone (N=123)
Anaemia (Blood and lymphatic system disorders) | 34 (53) | 40 (57)
Leukopenia (Blood and lymphatic system disorders) | 10 (21) | 9 (16)
Neutropenia (Blood and lymphatic system disorders) | 49 (120) | 33 (63)
Thrombocytopenia (Blood and lymphatic system disorders) | 26 (49) | 19 (27)
Constipation (Gastrointestinal disorders) | 30 (37) | 26 (27)
Diarrhoea (Gastrointestinal disorders) | 21 (30) | 27 (35)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 7 (7)
Nausea (Gastrointestinal disorders) | 23 (26) | 16 (19)
Vomiting (Gastrointestinal disorders) | 10 (17) | 13 (14)
Asthenia (General disorders) | 15 (21) | 14 (17)
Chest pain (General disorders) | 9 (11) | 5 (6)
Fatigue (General disorders) | 33 (36) | 37 (44)
Oedema peripheral (General disorders) | 22 (25) | 20 (23)
Pyrexia (General disorders) | 26 (35) | 19 (23)
Alanine aminotransferase increased (Investigations) | 10 (11) | 4 (4)
Blood creatinine increased (Investigations) | 7 (10) | 4 (4)
Neutrophil count decreased (Investigations) | 16 (28) | 17 (26)
Platelet count decreased (Investigations) | 7 (11) | 10 (12)
Weight decreased (Investigations) | 7 (7) | 5 (5)
White blood cell count decreased (Investigations) | 13 (19) | 11 (21)
Decreased appetite (Metabolism and nutrition disorders) | 9 (9) | 8 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (7) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 11 (16) | 8 (9)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (6) | 8 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (11) | 16 (17)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (15) | 21 (23)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15 (16) | 14 (15)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 (10) | 11 (13)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 12 (14) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (8) | 7 (7)
Dizziness (Nervous system disorders) | 16 (19) | 14 (15)
Headache (Nervous system disorders) | 16 (20) | 5 (7)
Neuropathy peripheral (Nervous system disorders) | 8 (8) | 5 (5)
Tremor (Nervous system disorders) | 10 (11) | 10 (10)
Depression (Psychiatric disorders) | 7 (7) | 3 (3)
Insomnia (Psychiatric disorders) | 10 (11) | 17 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (23) | 18 (21)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 (26) | 19 (25)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 3 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 10 (10)
Rash (Skin and subcutaneous tissue disorders) | 12 (13) | 10 (12)
Nasopharyngitis (Infections and infestations) | 7 (7) | 6 (8)
Pneumonia (Infections and infestations) | 7 (7) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 21 (27) | 25 (33)
Urinary tract infection (Infections and infestations) | 1 (1) | 8 (9)

LIMITATIONS AND CAVEATS:
The MK-3475-183 study was stopped/terminated early. Endpoint statistics may be biased due to the incomplete treatment and follow-up of participants after study termination

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/77/NCT02576977/Prot_SAP_001.pdf